CLINICAL TRIAL: NCT02391766
Title: Psychosocial Group Intervention to Enhance Empowerment of People With Dementia and Their Caregivers: Study Protocol for a Randomized Controlled Trial
Brief Title: Group Intervention Empowerment Dementia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: Principal Investigator, daniel serrani, PROFESSOR, Universidad Nacional de Rosario
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PGIED01; ´GIED01 (Registry Identifier: PGIED01)
Record Dates: First submitted 2014-02-04; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Empowerment; Self Efficacy; Quality of Life
Keywords: Self-management; Caregiving; Quality of life; Empowerment
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- empowerment group (Active Comparator): empowerment intervention by us for us guides
  Interventions: Behavioral: empowerment
- no treatment group (Placebo Comparator): dementia patients treatment as usual
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: empowerment — The groups of 10 participants meet once a week for eight weeks. last for four hours
  topics on dementia and prevention of further cognitive decline, active lifestyle and emotional well-being, spousal relationship, future planning kinds of active learning used are working in pairs and brainstorming sessions.
  Other Names: by us for us guides
  Arms: empowerment group
Behavioral: usual care
  Arms: no treatment group

SUMMARY:
After diagnosis of a dementing illness, patients and their spouses have many concerns related to the disease and their future. This often leads to poor psychological well-being and reduced health-related quality of life (HRQoL) of the family. Support for Empowerment has been proven to be an effective method to improve prognosis of asthma, heart failure, osteoarthritis.and diabetes. However empowering interventions have not been studied in dementia. Therefore, the investigators aim was to examine, in an objective-oriented group intervention, the efficacy of empowerment support program (ESP) on the HRQoL of dementia patients and their spousal caregivers as well as on the sense of competence and psychological well-being of caregivers.

Methods: During the years 2014 to 15, 180 dementia patients and their spouses will be recruited from memory clinics or day centers and randomized into two arms: 90 patients for group-based ESP sessions including topics selected by the participants and the use of the by us for us guides, 90 patients will serve as controls in usual community care. Sessions may include topics on dementia, active lifestyle and prevention for cognitive decline, spousal relationship, future planning and emotional well-being. The patients and spouses will have their separate group sessions (ten participants per group) once a week for eight weeks.

DETAILED DESCRIPTION:
Diagnoses and medications are confirmed from medical records provided by the couples. Charlson's comorbidity index is calculated to assess the severity and prognostic value of the participants' disease burden . Health-related quality of life (HRQoL) of the patients is assessed by using the 15D instrument Dementia patients are also assessed with the Clinical Dementia Rating Scale (CDR) the Mini Mental State Examination (MMSE) Other measurements include activities of daily living (ADL), instrumental activities of daily living (IADL) The presence of advance directives, such as a living will, are inquired about. Clinical measurements include height, weight, blood pressure and hand grip strength. The spousal caregivers are asked questions concerning the impact of their spouse's dementia diagnosis and they are assessed by the RAND-36 HRQoL instrument, 12-item General Health Questionnaire (GHQ-12) the Center for Epidemiologic Studies Depression Scale (CES-D) the randomization is performed by telephone to a randomization center. Couples are randomly allocated by means of computer-generated random numbers. Every randomization result will appear in the program after the participants name has been written and the person executing the randomization has confirmed the process with her initials. Participating couples are assessed by two study nurses three times over nine months: at baseline, three, and nine months. Use of health services, institutionalizations and mortality of both patients and caregivers will be retrieved from the central registers until 24 months from the baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* patients with dementia
* home dwelling with spouse
* not in the terminal phase of illness (estimated prognosis > one year)
* able to move independently (with or without devise)
* no severe hearing loss

Exclusion criteria:

* neurological disease
* other medical conditions
* head trauma
* inability to move independently

Ages: 56 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
patients' HRQoL (15D) | 8 weeks
  patients' HRQoL (15D)

SECONDARY OUTCOMES:
caregivers' psychological well-being (GHQ-12) | 8 weeks
  caregivers' psychological well-being (GHQ-12)
caregivers sense of competence (SCQ). | 8 weeks
  sense of self fulfillment and accomplishment in providing care to dementia patients
spousal caregivers' HRQoL (RAND-36) | 8 weeks
  spousal caregivers' HRQoL (RAND-36)

CONTACTS AND LOCATIONS:
Overall Officials: daniel serrani, Principal Investigator — Universidad Nacional de Rosario
Locations (1):
- Faculty of Psychology, Rosario, Santa Fe Province, Argentina